CLINICAL TRIAL: NCT04297644
Title: A Single-Center, Prospective Pilot Study to Verify the Algorithm of mCVI® to Accurately Capture Pulse Rate and Respiratory Rate in 10 Healthy Subjects in Comparison to Commercially-Available Masimo Pulse Oximeter Devices
Brief Title: mCVI Pilot Study: Algorithm Verification
Status: Completed | Type: Observational
Sponsor: Intelomed, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mCVI001
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Algorithm Verification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
This single center pilot study is to verify the algorithm of mCVI® to accurately capture pulse rate and respiratory rate in 10 healthy subjects in comparison to commercially-available Masimo pulse oximeter devices. This is a non significant risk device.

DETAILED DESCRIPTION:
In this pilot study the mCVI device is a mobile application used to simply verify the algorithm when the mobile video reads a patients pulse rate and respiratory rate while spontaneously breathing. There is no facial recognition technology. There is no immediate feedback given to the research team to act upon or provide for further clinical care decisions. In real time, the mCVI device will be compared to two commercially available pulse oximeter devices in a single visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients between the ages of 21 - 70

Exclusion Criteria:

* Medical conditions that could compromise a patient's ability to provide for all breathing samples, pedal the Cubii Pro elliptical, or follow instructions
* Medications that could compromise a patient's ability to participate in the study
* Documented medical history of respiratory or cardiovascular disease
* Excessive facial hair, facial deformities, or obstructions that could compromise the recording of pulse rate and respiratory rate of the mCVI®
* Missing digits or fingers on one or more hand that would prevent proper recording of Masimo pulse oximeter devices
* Patients wearing nail polish, acrylic nails, or rings on the ring finger of either hand that would prevent the proper use of Masimo pulse oximeter device
* Recent (≤ 1 month) surgical procedure of any kind
* Current participation in another investigational clinical trial
* Inability to provide informed consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 2 months
  To measure mCVI® respiration rate against Masimo pulse oximeter in people with different skin types.

SECONDARY OUTCOMES:
Secondary Objective | 2 months
  To measure mCVI® pulse rate against Masimo pulse oximeter in people with different skin types.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research South, INC, McMurray, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No